CLINICAL TRIAL: NCT03429569
Title: Comparison in Confocal Microscopy and Optical Coherence Tomography of Postoperative Morphological Changes of Keratoconus Treated by Cross-linking of Collagen in Accelerated Procedure and in Iontophoresis Procedure
Brief Title: Cross-Linking ACcéléré Iontophorèse Confocal kératocONE
Acronym: CLACICONE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-369; 2015-A00242-47 (Other: 2015-A00242-47)
Record Dates: First submitted 2017-11-28; First posted 2018-02-12 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Keratoconus
Keywords: Keratoconus; Cross-linking; Confocal microscopy; Postoperative morphological; Iotonphoresis
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accelerated conventional technique (Sham Comparator): Pachymetry greater than 400μm
  Topographic criteria for keratoconus evolution:
  Variation over a 6-month period of the following changes:
  An increase equal to or greater than 1D of maximum keratometry (Kmax) And / or an increase in mean keratometry (Kmean) greater than or equal to 0.75D And / or an increase in the difference between the meridian and the most arched and the least arched (Kmax-Kmin) greater than or equal to 0.75D And / or a decrease in the central thickness greater than or equal to 2% Criteria of non-inclusion Age under 18 Ectasies post LASIK Pregnant women breastfeeding Major corneal opacities Absence of consent to participation in the study No affiliation to Social Security or State Medical Aid (AME) or Universal Medical Coverage (CMU)
  Interventions: Drug: Cross linking
- iontophoresis (Sham Comparator): Pachymetry greater than 400μm
  Topographic criteria for keratoconus evolution:
  Variation over a 6-month period of the following changes:
  An increase equal to or greater than 1D of maximum keratometry (Kmax) And / or an increase in mean keratometry (Kmean) greater than or equal to 0.75D And / or an increase in the difference between the meridian and the most arched and the least arched (Kmax-Kmin) greater than or equal to 0.75D And / or a decrease in the central thickness greater than or equal to 2% Criteria of non-inclusion Age under 18 Ectasies post LASIK Pregnant women breastfeeding Major corneal opacities Absence of consent to participation in the study No affiliation to Social Security or State Medical Aid (AME) or Universal Medical Coverage (CMU)
  Interventions: Drug: Cross linking

INTERVENTIONS:
Drug: Cross linking — Accelerated cross-linking procedure: (Total duration: 40 minutes)

SUMMARY:
A monocentric, parallel-arm, prospective, randomized therapeutic trial that compares the efficacy of two curative keratoconus treatment techniques by cross-linking collagen (accelerated conventional technique or iontophoresis). The primary endpoint will be the depth of the demarcation line measured by confocal microscopy and OCT at 1 month. This line represents the limit depth between treated and untreated stroma.

DETAILED DESCRIPTION:
A two-arm, parallel, open-label, prospective, randomized therapeutic trial comparing two management strategies. The goal is to describe and compare, thanks to in vivo confocal microscopy and optical coherence tomography (OCT), the structural modifications observed postoperatively on evolutive keratoconus treated by cross-linking of collagen in accelerated procedure and iontophoresis. The study will be monocentric and will take place in the ophthalmology department of Clermont-Ferrand University Hospital. Patients will be recruited through consultation dedicated to keratoconus (The ophthalmology department of Clermont-Ferrand is one of the 9 French centers of expertise for this pathology). Inclusion will be offered to all patients over 18 years old who meet the scalability criteria and who will benefit from a cross-linking procedure. Blind randomization will be performed between iontophoresis and accelerated procedure. The dates of the visits will be fixed, with a preoperative evaluation, and a follow-up follow-up on 6 months with controls at 1 month, 3 months and 6 months. Confocal microscopy imaging and OCT will be performed during the preoperative visit and during visits at 1 month, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pachymetry greater than 400μm

Topographic criteria for keratoconus evolution:

Variation over a period of 6 months of the following parameters:

An increase equal to or greater than 1D of maximum keratometry (Kmax) And / or an increase in mean keratometry (Kmean) greater than or equal to 0.75D And / or an increase in the difference between the most arched and the least arched meridian (Kmax-Kmin) greater than or equal to 0.75D And / or a decrease in corneal central thickness greater than or equal to 2%

Exclusion Criteria:

Ectasies post LASIK Pregnant women breastfeeding Major corneal opacities Absence of consent to participate in the study No affiliation to social security or State Medical Aid (AME) or Universal Medical Coverage (CMU)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08-12 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
depth of the demarcation line | at one month
  depth of the demarcation line measured by confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric CHIAMBARETTA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France